CLINICAL TRIAL: NCT03227783
Title: The Effect of Transcranial Direct Current Stimulation (tDCS) on Depression in Parkinson's Disease
Brief Title: The Effect of Transcranial Direct Current Stimulation (tDCS) on Depression in PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Sangjin Kim, Professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-0051
Record Dates: First submitted 2017-07-17; First posted 2017-07-24 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel, Sham-controlled, single-blinded study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS (Active Comparator): * Constant weak electric currents through scalp via two electrodes will be delivered.
  * Current intensity: 2mA, 20min/day
  Interventions: Device: transcranial direct current stimulation (tDCS)
- Sham tDCS (Sham Comparator): * a 1 mA current, for 30 s giving an initial sensation of tDCS while minimizing stimulatory effects
  * Ramp up and ramp down was over 10 s. (Ref. Loo CK et al., Br J Psychiatry 2012;200:52-9)
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — tDCS is one of non-invasive brain stimulation. Constant, low current is delivered to the specific brain areas to change brain plasticity.

SUMMARY:
Depression is common in Parkinson's disease (PD), but the effective treatment is not established yet. tDCS is a non-invasive brain stimulation to modulate brain function. The tDCS on the depression in general population were already conducted, but not in PD. This study is to know whether transcranial direct current stimulation (tDCS) is effective for the treatment of depression in PD. Participant will be asked to visit three consecutive days for the non-invasive stimulation.

ELIGIBILITY:
Inclusion Criteria:

* UK Parkinson's disease brain bank criteria
* more than 19 years old
* Able to provide consent for the protocol
* Depression (based on DSM-IV criteria)

Exclusion Criteria:

* Dementia
* Unpredictable symptom fluctuations
* Contraindication to tDCS (i) irritations, cuts, lesions in the brain (ii) any preexisting unstable medical conditions, or conditions that may increase the risk of stimulation such as uncontrolled epilepsy (iii) history of severe cranial trauma with alteration of the cranial anatomy or metallic intracranial implants (iv) history of seizure
* Subjects without the capacity to give informed consent
* If participation in the study would, in the opinion of the investigators, cause undue risk or stress for reasons such as excessive fatigue, general frailty, or excessive apprehension

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
BDI score | (1) before the1st visit (within one month) (2) right after the 3rd tDCS (3) within one months after the 3rd tDCS
  The changes of Beck depression inventory after tDCS

SECONDARY OUTCOMES:
HDRS score | (1) before the 1st visit (within one month) (2) right after 3rd tDCS, within 24 hours (3) within one months after the 3rd tDCS
  The changes of Hamilton Depression Rating Scale after tDCS
MADRS score | (1) before the 1st visit (within one month) (2) right after the 3rd tDCS, within 24 hours (3) within one months after 3rd tDCS
  The changes of Mongomery-Asberg Depression Rating Scale after tDCS
resting state functional MRI | (1) before the 1st visit (within one month) (2) after the 3rd tDCS, within 24 hours (on the same day as the 3rd tDCS)
  The changes of resting state functional MRI after tDCS

CONTACTS AND LOCATIONS:
Overall Officials: Sang Jin Kim, MD, PhD, Principal Investigator — Inje University
Locations (1):
- Inje university, Busan Paik Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No